CLINICAL TRIAL: NCT06337877
Title: Assessment of Sedation Depth Using Processed EEG in ICU Patients With ARDS Receiving Neuromuscular Blockade: A Prospective Observational Study"
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, associated professor, Tepecik Training and Research Hospital
Other Study IDs: pEEG ARDS
Record Dates: First submitted 2024-03-17; First posted 2024-03-29 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Sedation Complication; Acute Respiratory Distress Syndrome Due to COVID-19; Anesthesia Awareness
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Depth of sedation monitoring — In the study, group rates of patient state index (PSI) [(below 25); (25-50); (51-75); (above 75)] will be determined within a 24-hour timeframe in patients undergoing therapeutic paralysis. The concordance between PSI rates* determined at baseline (time zero) and Richmond Agitation-Sedation Scale (RASS) [(between -4 and -5); (between -3 and -2); (equal to or greater than -1)] rates will be assessed. Suppression rate (SR) and electromyography (EMG) values will be obtained from patients, and significant differences among PSI groups [(below 25); (25-50); (51-75); (above 75)] in terms of these data will be examined. Additionally, changes in Propofol (mg/hour), Midazolam (mg/hour), Fentanyl (mg/hour), and Rocuronium (mg/hour) values will be analyzed for each time interval.

SUMMARY:
"In intensive care units, therapeutic paralysis has been a routine treatment method for many years in a select group of patients. Sufficient and appropriate sedation in patients undergoing therapeutic paralysis is crucial to prevent awareness and reduce the risk of excessive sedation. Both inadequate and excessive sedation levels can be highly detrimental to the patient. Clinical assessment may not always provide accurate information regarding sedation depth. Recently, the frequency and workload of therapeutic paralysis treatment in intensive care units have increased due to COVID-19 pneumonia. Therefore, the investigators believe that inadequate sedation may be common in these patients. Processed electroencephalogram parameters such as bispectral index or patient state index (PSI), routinely used in operating rooms and intensive care units, are commonly used to indicate sedation depth. In this study, the investigators aimed to determine sedation levels in patients during paralysis, assess the prevalence of inadequate or excessive sedation, and observe the doses of sedatives and analgesics used."

ELIGIBILITY:
Inclusion Criteria:

* "Patients aged 18 years and older who have received continuous neuromuscular blocking agents for at least 24 hours."

Exclusion Criteria:

1. Patients under 18 years of age,
2. pregnant individuals
3. trauma patients,
4. intracerebral pathology
5. major bleeding
6. central nervous system diseases,
7. pre-existing poor neurological condition before admission to the intensive care unit,
8. inability to document continuous neuromuscular blocking agent infusion for at least 24 hours."

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients who has ARDS
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
To determine the sedation levels of patients during paralysis | For patients undergoing therapeutic paralysis, over a 24-hour period,"
  "In the study, for patients undergoing therapeutic paralysis, routinely applied non-invasive patient state index (0-100) values will be recorded. These recorded values will be blindedly recorded from the clinician, who will not be alerted or intervene based on the values."
The prevalence of inadequate or excessive sedation, | For patients undergoing therapeutic paralysis, over a 24-hour period,"
  "In the study, for patients undergoing therapeutic paralysis, routinely applied non-invasive patient state index (0-100) values will be recorded. These recorded values will be blindedly recorded from the clinician, who will not be alerted or intervene based on the values."

SECONDARY OUTCOMES:
Evaluation of Concordance Between Richmond Agitation-Sedation Scale (RASS), | The assessment process conducted immediately before the application of paralysis."
  Evaluation of Concordance Between Richmond Agitation-Sedation Scale [(+4)- (-5)], a scale used in clinical assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aykut Saritaş, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided